CLINICAL TRIAL: NCT00661960
Title: A Pilot Project of Virologic, Pharmacologic and Immunologic Correlates of Gastrointestinal-Associated Lymphoid Tissue Immune Reconstitution Following Raltegravir Therapy
Brief Title: Pilot Project of Virologic and Immunologic Correlates of GALT Immune Reconstitution Following Raltegravir Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200715792
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: HIV Infections; AIDS
Keywords: HIV Positive; AIDS; Antiretroviral Therapy; Gastrointestinal-Associated Lymphoid Tissue; Immune Reconstitution; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; HIV Seropositivity | interventions — Raltegravir Potassium; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): HIV Negative volunteers
- 2 (Active Comparator): HIV-Positive volunteers taking raltegravir in combination with two other nucleoside reverse transcriptase inhibitors (NRTI) medications
  Interventions: Drug: raltegravir
- 3 (Active Comparator): HIV-Positive volunteers taking efavirenz or any other non-nucleoside reverse transcriptase inhibitors (NNRTI) in combination with two other nucleoside reverse transcriptase inhibitor (NRTI) medications
  Interventions: Drug: efavirenz

INTERVENTIONS:
Drug: raltegravir — 400mg tablet twice daily by mouth for nine months
  Other Names: Isentress
  Arms: 2
Drug: efavirenz — 600mg capsule once daily by mouth without regard to food
  Other Names: Sustiva
  Arms: 3

SUMMARY:
This research is being done to study how the immune system in the small intestine improves after taking antiretroviral (anti-HIV) medications. The main purpose is to measure the increase in the numbers of immune cells in the intestine to see if one type of HIV medication gives different results than other types of HIV medications.

DETAILED DESCRIPTION:
While the world-wide AIDS epidemic continues to impact millions of individuals, effective anti-HIV medications have substantially reduced morbidity and mortality for those patients able to adhere to combination regimens. Despite improved survival, durable virologic suppression, and increases in peripheral CD4+T-cell counts in patients receiving potent antiretroviral therapy (ART), immune reconstitution remains incomplete as measured by a number of additional surrogate markers. Perhaps critically important among areas of apparent incomplete immune recovery is the gastrointestinal-associated lymphoid tissue (GALT), where CD4+T-cells repopulate very slowly, if at all. Raltegravir is a new ART agent from a novel class of HIV inhibitors, integrase inhibitors, that results in rapid suppression of HIV and recovery of peripheral CD4+T-cells. This project proposes to examine whether volunteers receiving raltegravir recover GALT immune cells more completely than those taking comparator ART.

ELIGIBILITY:
Inclusion Criteria:

* willing to sign consent form
* no known GI pathology
* no anticipated antiretroviral therapy adjustments or changes
* males & females between the ages of 18 & 50 years
* no active opportunistic infections (OI) or therapy for OI within 30 days of entry
* can be on secondary prophylaxis with a history of AIDS defining illness
* per standard of care requirements, all females of child-bearing potential must agree to use barrier methods to prevent pregnancy or be abstinent from activity while on study

Exclusion Criteria:

* abnormal coagulation parameters (PT > or equal to 1.2 ULN)
* thrombocytopenia (platelet count < 50,000 within 6 weeks)
* contra-indications to upper endoscopy or conscious sedation
* anemia (> or equal to grade 1)
* aspirin, ibuprofen, warfarin or other agents that interfere with the coagulation cascade are prohibited within 1 week of endoscopy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2010-09 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Asmuth, M.D., Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - CARES Clinic, Sacramento, California
  - UC Davis Medical Center, Sacramento, California

REFERENCES:
- [Result] Asmuth DM, Ma ZM, Mann S, Knight TH, Yotter T, Albanese A, Melcher GP, Troia-Cancio P, Hayes T, Miller CJ, Pollard RB. Gastrointestinal-associated lymphoid tissue immune reconstitution in a randomized clinical trial of raltegravir versus non-nucleoside reverse transcriptase inhibitor-based regimens. AIDS. 2012 Aug 24;26(13):1625-34. doi: 10.1097/QAD.0b013e3283546595. PMID 22820612
- [Derived] Ellis CL, Ma ZM, Mann SK, Li CS, Wu J, Knight TH, Yotter T, Hayes TL, Maniar AH, Troia-Cancio PV, Overman HA, Torok NJ, Albanese A, Rutledge JC, Miller CJ, Pollard RB, Asmuth DM. Molecular characterization of stool microbiota in HIV-infected subjects by panbacterial and order-level 16S ribosomal DNA (rDNA) quantification and correlations with immune activation. J Acquir Immune Defic Syndr. 2011 Aug 15;57(5):363-70. doi: 10.1097/QAI.0b013e31821a603c. PMID 21436711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are recruited from the specialty clinic and their friends or family.
Pre-assignment Details: no special pre-assignment details
Groups:
- Negative Volunteers: HIV Negative volunteers
- HIV-postive Randomized to Raltegravir: HIV-Positive volunteers taking raltegravir in combination with two other nucleoside reverse transcriptase inhibitors (NRTI) medications
- HIV-postive Randomized to NNRTI: HIV-Positive volunteers taking efavirenz or any other non-nucleoside reverse transcriptase inhibitors (NNRTI) in combination with two other nucleoside reverse transcriptase inhibitor (NRTI) medications
Period: Overall Study
Arm/Group | Negative Volunteers | HIV-postive Randomized to Raltegravir | HIV-postive Randomized to NNRTI
Started | 5 | 10 | 10
Completed | 5 | 7 | 9
Not Completed | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Volunteers | HIV-postive Randomized to Raltegravir | HIV-postive Randomized to NNRTI | Total
Number analyzed (Participants) | 5 | 10 | 10 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 10 | 25
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (5) | 37 (5) | 45 (5) | 38 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 8
  Male | 4 | 6 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: the Percentage of CD3+/CD4+ Cells Per Cubic Millimeter at the Effector Sites in the Duodenal Tissues Obtained From Volunteers to the Antiretroviral Therapy Regimen Over Time.
Description: Duodenal tissue immune cell subsets were measured by flow cytometry.
Time Frame: nine months
Population: all subjects who completed all study visits
Measure: Median (Inter-Quartile Range); unit: % CD3/CD4 T-cells in GALT tissue
Arm/Group | Negative Volunteers | HIV-postive Randomized to Raltegravir | HIV-postive Randomized to NNRTI
Number analyzed (Participants) | 5 | 7 | 9
% CD3/CD4 T-cells in GALT tissue | 55.3 [42 to 67] | 11.7 [9.1 to 22.3] | 9.9 [8.7 to 18.2]

ADVERSE EVENTS:
Arm/Group | Negative Volunteers | HIV-postive Randomized to Raltegravir | HIV-postive Randomized to NNRTI
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Limitations of the study include small numbers of subjects over all - Several subjects dropped out due to moving out of the region and lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No